CLINICAL TRIAL: NCT05536765
Title: Augmented Reality-assisted Surgical Exposure of an Impacted Tooth
Brief Title: Augmented Reality in Oral Surgery
Status: Completed | Type: Observational
Sponsor: D'Albis Dental (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, Principal Investigator, D'Albis Dental
Other Study IDs: AR in Dentistry
Record Dates: First submitted 2022-09-06; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-06

CONDITIONS: Impacted Tooth
Keywords: Augmented reality; Oral Surgery; Computer guided surgery; Computer assisted surgery
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with impacted tooth
  Interventions: Procedure: Surgical exposure of impacted tooth

INTERVENTIONS:
Procedure: Surgical exposure of impacted tooth — The therapeutic approach of surgical exposure of impacted teeth is performed by preparing a flap and removing the cortical bone around the crown of the teeth.
  This procedure provides optimal conditions for the orthodontist. In fact, surgical exposure allows the orthodontist to bond the impacted tooth in the correct position depending on the intended direction to apply the correct traction forces for alignment.

SUMMARY:
A digital workflow was used to assist the oral surgeon in pre-orthodontic exposure of a vestibular impacted canine using Augmented Reality.

Through software for the Object Recognition and Tracking, the researchers expand reality with cone beam computer tomography digital contents to optimize the outcome of surgery. The real-time video frames of the operating field aligned with the three-dimension file of the impacted tooth, were used as a guide to evaluate the surgical access to perform a minimally invasive flap and osteotomy.

DETAILED DESCRIPTION:
This study evaluate an AR-assisted approach for surgical exposure of a maxillary impacted canine. The usual protocol is the following:

* Maxillary arches were scanned, and their occlusal relationship was registered using an optical intraoral scanner.The file was exported in Polygon File Format (PLY)
* Using open-source CAD software, the part of the upper arch was selected from the first premolar to the other first premolars The teeth, the incisal edges and the cusps of the anterior sector were the anatomical markers required to match the patient's mouth and perform the object recognition.To this file that corresponded faithfully to reality we added the digital information required, that is, the position of the impacted crown of the canine
* From the maxillary CBCT, DICOM files were imported in open-source medical software for segmentation and exportation of an STL file of the area of interest
* Two 3D files obtained were imported into a CAD-CAM design software for superimposition. 3D file consisting of the intraoral scan plus the endosseous position of the crown of the impacted canine was exported
* A full HD video camera was positioned in front of the patient's mouth, connected via an HDMI cable to a laptop
* The AR software was then started, and the video camera was associated as an input source The software recognizes edges of files in images transmitted from the camera and overlap the object to the video images.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an impacted tooth in aesthetic area
* Good health according to the System of the American Society of Anesthesiology
* No general medical contraindication for oral surgery
* Good periodontal health

Exclusion Criteria:

* Smoking more than 15 cigarettes a day • Untreated periodontitis
* Pregnancy
* Acute infections

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with impactet tooth. In growing age or not.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluation in mm of the superimposition between 3d model and patient anatomicals structures. | 1 month
  Evaluation of a software that uses algorithms to recognize and track 3D files in a real-time frame to visualize the endosseous position of the crown of an impacted tooth in order to plan the surgical exposure in a precise and minimally invasive manner. Evaluation through the software the distance in millimeters between the superimposition of the 3d model ed the patient's structures.

CONTACTS AND LOCATIONS:
Locations (1):
- Giuseppe D'Albis, Mola di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No